CLINICAL TRIAL: NCT06680804
Title: Factors Affecting Success of Vaginal Birth After Cesarean Section in Sohag University Hospitals
Brief Title: Factors Affecting Success of Vaginal Birth After Cesarean Section
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nahla Rashwan Ezz-eldine, Resident at obstetrics and gynecology , sohag university, Sohag University
Other Study IDs: soh-Ned-15-10_9MS
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Vaginal Delivery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Successful VBAC group: Successful VBAC group whose take chance for vaginal delivery.
  Interventions: Other: chance for vaginal delivery.
- Group II: Failed VBAC group: Failed VBAC group whose take chance for vaginal delivery.
  Interventions: Other: chance for vaginal delivery.

INTERVENTIONS:
Other: chance for vaginal delivery. — chance for vaginal delivery in patients who had delivered by Caesarean section in first pregnancy

SUMMARY:
Factors affecting Success of Vaginal Birth After Cesarean Section in Sohag University Hospitals

DETAILED DESCRIPTION:
* Clinical data will be collected from the participants including demographic details such as age, maternal age, parity, BMI, gestational age based on last menstrual period or early ultrasound scans available.
* Full medical and surgical history, previous CS details as an indication, and previous complications.
* Patients' clinical abdominal and per vaginal examination on admission (cervical dilatation, effacement head station, and position).
* CTG attached on admission (to exclude fetal distress).
* Laboratory investigations that will be done before delivery and postpartum, Labor progress on the partogram will be assessed as regard duration of both first and second stages of labor if any instrumental delivery will be done.
* Radiology investigations such as US.
* Records for patients' vital signs, fetal cardiac activity during labor, vaginal bleeding, delivery notes, fetal weight, and 5 minutes APGAR score, and any recorded maternal or fetal complications.
* If failed VBAC: Causes of failure maternal and fetal outcomes will be recorded and immediate CS to be done

ELIGIBILITY:
Inclusion Criteria:

* • Age from 20 to 40 years.

  * Time interval more than 1.5 years from previous caesarean section.
  * Single viable full-term pregnancy in vertex presentation.
  * Reactive cardiotocography (CTG) on admission.
  * Spontaneous labor onset.
  * Clinically adequate pelvis.
  * Single fetus
  * Average AFI fetus

Exclusion Criteria:

* • Women with previous upper segment cesarean section or hysterotomy scar.

  * Any obstetric complications such as fetal malpresentation, placenta previa, or medical disorders like diabetes mellitus or preeclampsia.
  * Presence of any signs and symptoms of scar dehiscence or ruptured uterus, known uterine fibroid or anomaly.
  * Suspected fetal macrosomia (weight more than 4 kg).
  * Multifetal pregnancy.
  * Parturient women who refused the trial of vaginal birth after caesarean section.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: All patients admitted for vaginal delivery with previous lower segment cesarean section . Age from 20 to 40 years.Time interval more than 1.5 years from previous caesarean section.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
successful vaginal delivery | From November 2024 to April 2025
  successful vaginal delivery in patients who had delivered by Caesarean section in first pregnancy

IPD SHARING:
Plan to Share IPD: No